CLINICAL TRIAL: NCT06517927
Title: Prevalence of Long-term Dental Effects of Chemotherapy in Childhood Cancer Survivors Diagnosed With Cancer Before the Age of 10
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DENTAL CHEMO
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Chemotherapy Effect; Dental Caries; Malocclusion; Childhood Cancer; Tooth Defect
Keywords: Childhood cancer survivors; Dental defect
MeSH Terms: conditions — Dental Caries; Malocclusion; Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventionnal study, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer survivor (Experimental)
  Interventions: Diagnostic Test: Clinical and radiographic dental examination
- Control (Active Comparator)
  Interventions: Diagnostic Test: Clinical and radiographic dental examination

INTERVENTIONS:
Diagnostic Test: Clinical and radiographic dental examination — complete clinical oral examination + intra-oral and panoramic x-rays

SUMMARY:
To date, there are no methods for assessing the risk of oral developmental defects that could predict long-term adverse effects in childhood cancer survivors. Having such a method at our disposal would enable us to better assess the risk to develop those defects and will help us provide new prevention and treatment strategies to ensure a healthy oral development.

The aims of this study are :

* Assess the caries risk in childhood cancer survivors compared with a control group.
* Assess the dental development defects risk in childhood cancer survivors compared with a control group.

DETAILED DESCRIPTION:
This will be an international study comparing the Childhood Cancer Survivors (CCS) and a control group.

A questionnaire will be provided to the patients to gather information. A standard of care dental examination will then take place in a dental office in the Cliniques Universitaires Saint-Luc. We also collect medical data to complete the files.

ELIGIBILITY:
Inclusion Criteria:

* age below 10 at cancer diagnosis (for the CCS group).
* Chemotherapy must have been used to treat the patient (For the CCS group).
* The patient is 12 years old or older at the time of the follow-up appointment of the present study

Exclusion Criteria:

* A patient who was diagnosed and treated after 10 years old.
* Patient below 12 years old at time of study recruitment
* Patients with syndrome or diseases that involve teeth impairment*
* Pregnant patient
* Refusal or inaptitude to undergo dental and radiographic examination

Ages: 12 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of the caries experience by using the Decay Missing Filled Teeth score (DMFT) | Thoughout the entire study, approximately during 2 years
  Assess the impact of the chemotherapy agents on the risk of ulterior caries development

SECONDARY OUTCOMES:
Assessment of the prevalence of dental development defects (DDD) | Thoughout the entire study, approximately during 2 years
  Assess the impact of the chemotherapy agents on the risk of ulterior dental development defect

CONTACTS AND LOCATIONS:
Overall Officials: Maëlle De Ville de Goyet, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No